CLINICAL TRIAL: NCT02328248
Title: Randomized Control Trial (RCT) That the Usage With Biological Patch Versus Plastic in the Laparoscopic Repair
Brief Title: Usage of Biological Patch Versus Plastic in the Laparoscopic Repair of Hiatal Hernias
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Xiaonan Liu, associate professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HH-001
Record Dates: First submitted 2014-11-28; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Hiatal Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biological patch (Experimental): Use biological patch (Biodesign Surgisis Tissue Graft from Cook Biotech Incorporated) to repair hiatal hernia laparoscopically
  Interventions: Procedure: Biological patch
- Plastic patch (Placebo Comparator): Use plastic patch (Parietex Composite from Sofradim Production) to repair hiatal hernia laparoscopically

INTERVENTIONS:
Procedure: Biological patch — Use biological patch as opposed to plastic patch to repair hiatal hernia laparoscopically
  Arms: Biological patch

SUMMARY:
The purpose of this study is to observe the effective and safety in the laparoscopic repair of hiatal hernia using biological patch versus plastic.

DETAILED DESCRIPTION:
observation indicator:

1. incidence rate of complications,
2. postoperative hospital stay
3. readmission rate in 1st month after operation
4. recurrence rate after operation
5. hospitalization costs
6. Self-evaluation of gastroesophageal reflux symptoms and quality of life(QOL) in 6th-month, 1st-year,2nd-year,3rd-year,4th-year and 5th-year after operation

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Hiatal hernia
* Consistent with operation indications throughout the guideline of hiatal hernia by the Chinese Medical Association in 2003
* randomly select patch agreed by patients and family members

Exclusion Criteria:

* Poor general condition
* severe organ dysfunction
* No-tolerate anesthesia
* No-suitable for operation
* Emergency operation needed
* Serious adverse events appeared during the operation
* Sever intraperitoneal adhesion existed
* glucocorticoid with long-term use
* immunocompromised patients
* spirit disease patients
* automatically exit
* women who pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of complications in all case | five years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Liu, Ph.D, Study Chair — Xijing Hospital